CLINICAL TRIAL: NCT06694064
Title: Evaluation of Mineral Trioxide Aggregates and Grape Seeds Extract Effectiveness in Pulpotomy of Primary Molars
Brief Title: Evaluation of Mineral Trioxide Aggregates and Grape Seeds Extract Effect on Pulpotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, sara nabil, Associate Professor of pediatric dentistry, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC- PD-23-01
Record Dates: First submitted 2024-10-21; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — Pulpotomy; Histological Techniques

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mta group (Experimental): after pulpotomy the pulp stumps subgected to mta material
  Interventions: Procedure: Pulpotomy; Procedure: extraction for histologic examination
- Grape seed group (Experimental): after pulpotomy the pulp stumps subjected to grape seed
  Interventions: Procedure: Pulpotomy; Procedure: extraction for histologic examination

INTERVENTIONS:
Procedure: Pulpotomy — Pulpotomy will be done for mta group
Procedure: extraction for histologic examination — after pulp therapy the teeth exrtracted for histologic examination

SUMMARY:
Pediatric dentistry has always debated the benefits of vital pulp therapy. AIM: The current study was done to differentiate the histo-pathological findings of MTA versus grape seed extract in primary teeth undergoing pulpotomy as pulp dressing substances. Materials and Methods: According to the inclusion criteria, 16 primary teeth were selected in each group. Randomly and equally, the teeth were split into two groups: (MTA group) Group I, and (GSE group) Group II. After nine months, under a light microscope the teeth were evaluated and a clinical follow-up was conducted. Periapical radiographs were also taken at this time.

ELIGIBILITY:
Inclusion Criteria:

* healthy patients with carious primary molars

Exclusion Criteria:

* root resorption

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-09-02 (Actual)

PRIMARY OUTCOMES:
evaluate pain of the teeth | 6 months
  The lack of any clinical indications of pulp degeneration, such as the history of spontaneous pain, pain on percussion, swelling, pathological mobility, or sinus tract

SECONDARY OUTCOMES:
absence of radiolucency | 6 months
  No signs of periapical orfurcal radiolucency, widening of the periodontal ligament (PDL), or pathological root resorption (internal or external).

CONTACTS AND LOCATIONS:
Locations (1):
- Alazhar University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Individual Participant Data Set — https://pubmed.ncbi.nlm.nih.gov/36464977/